CLINICAL TRIAL: NCT01523509
Title: The Use of Radiographic Contrast to Differentiate Cavitated From Non-cavitated Dental Caries
Brief Title: Use of Radiographic Contrast to Detect Dental Caries
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Douglas K Benn DDS, PhD, Professor and PI, Creighton University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CU IRB-01
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Dental Caries
Keywords: Dental Caries; Radiography, Dental; Contrast media; Tooth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contrast (Experimental): All subjects will be in one group who will have a control radiograph of teeth before applying the Sodium Iodide contrast agent topically between the teeth (the intervention) when another radiograph will be taken to test for the presence of contrast in a cavity.
  Interventions: Device: Radiographic contrast agent. Sodium Iodide.

INTERVENTIONS:
Device: Radiographic contrast agent. Sodium Iodide. — Application of Sodium Iodide contrast topically to tooth immediately followed by radiograph.

SUMMARY:
The proposed test is intended to enable dentists to differentiate between cavitated and non-cavitated tooth decay in the areas where teeth are in contact (interproximal surfaces). In these areas, dentists cannot visually inspect for caries, and currently bitewing X-rays (BWs) only correctly detect the presence of enamel decay 15-25% of the time. This low sensitivity can lead to late treatment resulting in unnecessarily large fillings, crowns, pain, root canals, and possible later loss of teeth.

Hypothesis: Use of radiographic contrast on teeth will increase the accuracy of detection of early cavitation from 58% to 90%.

DETAILED DESCRIPTION:
Tooth sites will be recorded by tooth number, type of surface (mesial, distal,occlusal), cavitated, non-cavitated, healthy. Radiographs will similarly be scored.Although contrast agents are classified as drugs this is not a study of drug properties or effect on cells since the properties of the agent are already well know and its safety record well established. This study will be recording the radiopacity of the contrast agent on healthy tooth surfaces, non-cavitated tooth surfaces and cavitated tooth surfaces. The outcome for each surface type will be presence or absence of a radiopacity on a radiograph which will be made at the one and only visit for each study subject. The radiograph contains the data from the intervention (placement of contrast agent) and the outcome will be assessed some weeks later after the completion of the data collection.

ELIGIBILITY:
Inclusion Criteria:

* must have a minimum of 2 adjacent teeth so that interproximal surfaces of interest are in contact and hidden from direct visual inspection.
* the occlusal plane should be normal so that the interproximal contact regions are normal.
* English or Spanish speaker.

Exclusion Criteria:

* pregnant women
* a person who has participated in a similar study involving dental radiography within the last 12 months.
* fillings must not be present in the regions of interest.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Presence of a radiopacity below the tooth surface at a site likely to develop tooth decay. | Immediately after application of contrast agent.
  The PI will perform the clinical application of the contrast agent and radiograph the subject. In this way it will be known that the data has been collected. At a later date 3 independent dentists will be provided with blinded radiographs in a randomized order to report the presence or absence of cavitated caries lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas K Benn, DDS PhD, Principal Investigator — Creighton University
Locations (1):
- Creighton University School of Dentistry, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Benn DK, Cooper RL, Nunn ME, Edwards SE, Rocha-Sanchez SM. A radiographic method for distinguishing noncavitated from cavitated proximal carious lesions: A proof of concept clinical trial. Oral Surg Oral Med Oral Pathol Oral Radiol. 2021 Dec;132(6):715-726. doi: 10.1016/j.oooo.2021.02.014. Epub 2021 Feb 23. PMID 34083157